CLINICAL TRIAL: NCT03129191
Title: Audiological Benefit With Non-implantable Bone Conduction Hearing Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRL-NIBCH
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Hearing Loss, Conductive
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB arm (Active Comparator): Sequence:
  1. Aided with non-invasive bone conduction hearing aid A
  2. Aided with non-invasive bone conduction hearing aid B
  Interventions: Device: Non-invasive bone conduction hearing aid A; Device: Non-invasive bone conduction hearing aid B
- BA arm (Active Comparator): Sequence:
  1. Aided with non-invasive bone conduction hearing aid B
  2. Aided with non-invasive bone conduction hearing aid A
  Interventions: Device: Non-invasive bone conduction hearing aid A; Device: Non-invasive bone conduction hearing aid B

INTERVENTIONS:
Device: Non-invasive bone conduction hearing aid A — The intervention is a non-invasive bone conduction hearing device which is retained on the patient's head with an elastic headband.
Device: Non-invasive bone conduction hearing aid B — The intervention is a non-invasive bone conduction hearing device which is retained on the patient's head with an adhesive adapter that is placed behind the auricle.

SUMMARY:
Recently, a new non-invasive bone conduction hearing aid was introduced. The system is connected directly to the skin with an adhesive adapter to transmit the sound to the inner ear through bone vibrations. The objective of this study is to evaluate and compare the audiological benefit of the new bone conduction hearing aid and compare it to an existing bone conduction hearing aid in normal hearing adults with bilateral simulated conductive hearing loss.

An evaluation of the improvement on speech understanding in noise and sound localization allows to estimate the system performance and enables to derive recommendations for clinical usage of the novel hearing system. It is hypothesized that in the bilateral condition similar speech understanding in noise and sound localization performance can be achieved with the new system compared to existing bone conduction hearing aids that are pressed against the skull using a soft band.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults (age ≥ 18 years on the test date)
* Normal hearing thresholds (AC/BC-thresholds ≤ 20 dB HL, 0.25 to 8 kHz)
* German native speakers
* Willingness and ability to perform all tests required for the study

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Allergy against silicon (ear mold casting mass)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold in noise (S0NDIFF) | Day 1
  Speech reception threshold in noise (in dB SNR) measured with speech presented from the front (0° azimuth) and approximated diffuse noise presented from 4 speakers.

SECONDARY OUTCOMES:
Speech reception threshold in noise (S90NDIFF) | Day 1
  Speech reception threshold in noise (in dB SNR) measured with speech presented from the right side (90° azimuth) and approximated diffuse noise presented from 4 speakers.
Speech reception threshold in noise (S270NDIFF) | Day 1
  Speech reception threshold in noise (in dB SNR) measured with speech presented from the left side (270° azimuth) and approximated diffuse noise presented from 4 speakers.
Sound localization | Day 1
  Mean absolute localization error (in degrees)
Subjective evaluation of the sound quality | Day 1
  Assessment of the sound quality with questionnaire by Gabrielsson et al.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kompis, Prof, Principal Investigator — University Hospital Bern, Inselsptial
Locations (1):
- Hearing Research Laboratory, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided